CLINICAL TRIAL: NCT01774643
Title: A Feasibility Study Of Developing Murine Primary Xenografts From Biopsies Of Liver Metastases In Patients With Advanced Pancreatic Cancer
Brief Title: A Study of Pancreatic Cancer in Xenografts From Liver Metastases
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: XENO-METPANC
Record Dates: First submitted 2013-01-22; First posted 2013-01-24 (Estimated); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Cancer; Liver Metastases; Tumor Tissue Biopsy; Blood Samples
Keywords: Pancreatic cancer; Liver metastases; Tumor tissue biopsy; Blood samples; Xenografts; Murine; Genomic profiling; Circulating biomarkers
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatic cancer with liver metastases: Tumor tissue biopsy, blood samples

SUMMARY:
This is a feasibility study to perform image-guided liver biopsies in 25 patients who have pancreatic cancer with liver metastasis (cancer in the pancreas that has spread to the liver). This will contribute with samples for the bio-bank (bank of tumors) and develop xenografts (human tumors growing in mice) for further analysis of genes.

DETAILED DESCRIPTION:
This study might bring a better understanding of the metastatic pancreatic cancer and evaluate the differences between the metastatic and the primary pancreatic cancer (the type that does not have metastasis).

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 18 years old
* Pancreatic cancer with liver metastasis
* No contraindication to image-guided biopsy of liver metastasis, including uncontrolled bleeding diathesis, uncontrolled malignant pain, inability to lie supine etc) and no significant hepatic dysfunction.
* Provide written informed consent
* ECOG 0,1 or 2

Exclusion Criteria:

* Inability to lie supine for more than 30 minutes
* ECOG 3 or more
* Serious medical risk factors involving any of the major organ systems or including uncontrolled bleeding diathesis, uncontrolled malignant pain, inability to lie supine etc) and no significant hepatic dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer patients with liver metastases
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2013-01; Primary Completion 2015-04 (Actual); Study Completion 2022-11 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse events due to biopsies | up to 2 years
  Monitoring adverse events during trial related to biopsies
Number of successful xenografts | up to 2 years
  determine the "take rate" or success of establishing xenografts
Number of similarities and differences between original patient tumor sample with xenograft sample | up to 2 years
  complete histological and molecular comparison of original patient sample with murine xenograft
Engraftment rate compared to clinical data (response to treatment, disease-free survival, overall survival) | up to date of death from any cause
  determine the correlation between engraftment rate and clinical data (response to treatment, disease-free survival, overall survival).

CONTACTS AND LOCATIONS:
Overall Officials: Neesha Dhani, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada